CLINICAL TRIAL: NCT01449279
Title: A Pilot Study of Ipilimumab in Subjects With Stage IV Melanoma Receiving Palliative Radiation Therapy
Brief Title: Pilot Ipilimumab in Stage IV Melanoma Receiving Palliative Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Susan Knox, Associate Professor of Radiation Oncology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21970; SU-08242011-8306 (Other: Stanford University); MEL0005 (Other: OnCore)
Record Dates: First submitted 2011-10-05; First posted 2011-10-10 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipilimumab Treatment + Radiation Therapy (Experimental): Ipilimumab (BMS-734016, MDX010, MDX-CTLA4, Yervoy) will be administered as standard of care with base dose of 3 mg/kg iv over approximately 90 minutes every 3 weeks for a total of 4 treatments. Palliative radiation therapy to 1 to 2 sites of disease will start within 5 days of the first ipilimumab dose. Subjects will have follow up visits 2 to 4 weeks after the last ipilimumab dose and then every 3 months (±2 weeks) thereafter until progression of disease.
  Interventions: Drug: Ipilimumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab will be administered as a single agent standard of care with base dose of 3 mg/kg iv over approximately 90 minutes every 3 weeks for a total of 4 treatments.
  Other Names: MDX-101; Yervoy
Radiation: Radiation Therapy — Standard of care palliative radiation therapy will start within 5 days of the first ipilimumab dose. Dose is dependent upon lesion size and is determined by the radiation oncologist.
  Other Names: radiotherapy; radiation oncology

SUMMARY:
To determine the safety of local palliative radiation therapy used in combination with anti-CTLA-4 immunotherapy.

DETAILED DESCRIPTION:
This is a single institution, open-label, pilot study of palliative radiation therapy (RT) combined with ipilimumab in patients with stage IV melanoma. The primary objective of this study is to assess the safety of combining ipilimumab with palliative RT in patients with Stage IV melanoma. Secondary objectives are a) to assess the induction of anti-melanoma immune responses using laboratory correlative studies of T cell responses to melanoma antigens, and b) to compare tumor response rates and duration of response at unirradiated sites with responses in patients with Stage IV disease treated with ipilimumab alone on expanded access study CA184045. In this study, ipilimumab will be administered as recently approved by the FDA (3 mg/kg iv every 3 weeks for a total of 4 treatments). Palliative RT will start within 2 days of the first ipilimumab dose. Patients will be seen at least every 12 weeks for follow-up following completion of ipilimumab therapy until progression of disease by imaging criteria or increased symptomatology that requires another therapy. A total of 20 patients with previously treated unresectable metastatic melanoma requiring palliative radiation therapy will be treated on this pilot study over approximately 18 months. All subjects who receive study drug will be monitored for safety. Relevant tumor imaging studies will be obtained at baseline, 2-4 weeks following the 4th/last dose of ipilimumab, and then every 12 weeks until disease progression. This study will provide the safety data (and possibly early efficacy signals) needed to proceed with a randomized Phase II study for proof of principle. If compelling data is obtained supporting this IT + RT vaccine strategy, this approach will be extended to other solid tumor types.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   Before any study procedures are performed, subjects (or their legally acceptable representatives) will have the details of the study described to them, and they will be given a written informed consent document to read. Then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel.
2. Target Population

   * Histologically confirmed Stage IV melanoma.
   * Must have failed at least one systemic therapy for malignant melanoma or be intolerant to at least one prior systemic treatment.
   * Subjects with asymptomatic brain metastases are eligible. (Systemic steroids should be avoided if possible, or the subject should be stable on the lowest clinically effective dose, as steroids as they may interfere with the activity of ipilimumab if administered at the time of the first ipilimumab dose.)
   * Primary ocular and mucosal melanomas are allowed.
   * Must be at least 28 days since treatment with chemotherapy, biochemotherapy, surgery, radiation, or immunotherapy, and recovered from any clinically significant toxicity experienced during treatment.
   * Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
   * Life expectancy of ≥ 16 weeks.
   * Subjects must have baseline (screening/baseline) radiographic images, (e.g. brain, chest, abdomen, pelvis, and bone scans with specific imaging tests to be determined by the attending physician) within 6 weeks of initiation of ipilimumab.
   * Required values for initial laboratory tests:

     * White blood cell (WBC) ≥ 2000/uL (~ 2 x 10^9/L)
     * Absolute neutrophil count (ANC) ≥ 1000/uL (~ 1 x 10^9/L)
     * Platelets ≥ 75 x 10^3/uL (~ 75 x 10^9/L)
     * Hemoglobin ≥ 9 g/dL (~ 80 g/L; may be transfused)
     * Creatinine ~ 2 x upper limit of normal (ULN)
     * Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ~ 2.5 x ULN for subjects without liver metastasis ~ 5 times for liver metastases
   * Bilirubin: ~ 2.0 x ULN (except for subjects with Gilbert's Syndrome, who must have a total bilirubin of < 3.0 mg/dL)
   * No active or chronic infection with HIV, Hepatitis B, or Hepatitis C.
   * Two or more measurable sites of disease (≥ 1.5 cm) which include the disease site that requires palliative radiation therapy as well as ≥ 1 other disease site outside of the planned radiation therapy field.
3. Age and Sex

   * Men and women, at least 18 years of age.
   * Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study [and for up to 26 weeks after the last dose of investigational product] in such a manner that the risk of pregnancy is minimized.
   * WOCBP include any female who has experienced menarche and who has undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Post-menopausal is defined as:

     * Amenorrhea ≥ 12 consecutive months without another cause, or
     * For women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
   * Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of investigational product.

     c) Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last dose of investigational product] in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

1. Sex and Reproductive Status

   * WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study and for up to 8 weeks after the last dose of investigational product.
   * WOCBP using a prohibited contraceptive method.
   * Women who are pregnant or breastfeeding.
   * Women with a positive pregnancy test on enrollment or before investigational product administration.
2. Target Disease Exceptions

   * Subjects on any other systemic therapy for cancer, including any other experimental treatment.
   * Prior treatment with an anti-CTLA-4 antibody if treatment failure was due to adverse events (AEs). If a subject was discontinued from the prior anti-CTLA-4 treatment due to an AE or serious adverse event (SAE), regardless of the type of event, that discontinuation constitutes an exclusion criterion. If AEs were serious enough to require a subject's withdrawal from prior treatment, the subject should be excluded from this study.
   * A history of AEs with prior IL-2 or Interferon will not preclude subjects from entering the current study.
   * Subjects who relapsed in study MDX010-16 are not eligible for this study.
3. Medical History and Concurrent Diseases

   * Autoimmune disease: subjects with a documented history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease are excluded from this study as are subjects with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma]; systemic lupus erythematosus (SLE); autoimmune vasculitis [eg, Wegener's Granulomatosis]). Subjects with motor neuropathy considered of autoimmune origin (eg, Guillain-Barre Syndrome and Myasthenia Gravis) are excluded from this study.
   * Any subject who has a life-threatening condition that requires high-dose immunosuppressant(s)
   * Presence of known Hepatitis B or Hepatitis C infection, regardless of control on antiviral therapy
   * Subjects with melanoma who have another active, concurrent, malignant disease are not eligible for the CA184045 study, with the exception of subjects with adequately treated basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix.
4. Medical History and Concurrent Diseases

   * Prisoners or subjects who are involuntarily incarcerated.
   * Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
   * Any underlying medical or psychiatric condition that, in the opinion of the investigator, could make the administration of ipilimumab hazardous or could obscure the interpretation of adverse events.
   * Any non-oncology vaccine therapy used for prevention of infectious diseases for up to 4 weeks before or after any dose of ipilimumab, with the exceptions of amantadine and flumadine.
   * Central nervous system (CNS) metastases that require palliative radiation therapy; prior brain irradiation is allowed providing CNS disease is stable.
5. Additional Concomitant Treatments

   * Any investigational agents
   * Any other (non-CA184045 related) CTLA-4 inhibitors or agonists
   * CD137 agonists
   * Immunosuppressive agents (unless required for treating potential AEs)
   * Chronic systemic corticosteroids (unless required for treating treatment emergent AEs or required for management of signs or symptoms due to brain metastases, upon discussion with BMS medical monitor).

Eligibility criteria for this study have been carefully considered to ensure the safety of the study subjects and to ensure that the results of the study can be used. It is imperative that subjects fully meet all eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Knox, PhD, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hiniker SM, Reddy SA, Maecker HT, Subrahmanyam PB, Rosenberg-Hasson Y, Swetter SM, Saha S, Shura L, Knox SJ. A Prospective Clinical Trial Combining Radiation Therapy With Systemic Immunotherapy in Metastatic Melanoma. Int J Radiat Oncol Biol Phys. 2016 Nov 1;96(3):578-88. doi: 10.1016/j.ijrobp.2016.07.005. Epub 2016 Jul 15. PMID 27681753

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited during clinic visits at the Stanford Cancer Center clinic. Subjects were informed of all options and given time to ask questions before signing consent in a private room.
Groups:
- Ipilimumab Treatment + Radiation Therapy: Ipilimumab (BMS-734016, MDX010, MDX-CTLA4, Yervoy) will be administered as standard of care with base dose of 3 mg/kg iv over approximately 90 minutes every 3 weeks for a total of 4 treatments. Palliative radiation therapy to 1-2 sites of disease will start within 5 days of the first ipilimumab dose. Subjects will have follow up visits 2-4 weeks after the last ipilimumab dose and then every 3 months (±2 weeks) thereafter until progression of disease.
  Ipilimumab: Ipilimumab will be administered as a single agent standard of care with base dose of 3 mg/kg iv over approximately 90 minutes every 3 weeks for a total of 4 treatments.
  Radiation Therapy: Standard of care palliative radiation therapy will start within 5 days of the first ipilimumab dose. Dose is dependent upon lesion size and is determined by the radiation oncologist.
Period: Overall Study
Arm/Group | Ipilimumab Treatment + Radiation Therapy
Started | 22
Completed | 15
Not Completed | 7
Not completed — Lack of Efficacy | 5
Not completed — Toxicity | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab Treatment + Radiation Therapy
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: Years] | 59 [18 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Safety Measurement - Percentage of Patients Experiencing Serious Adverse Events (SAEs) in the First 4 Months of Treatment.
Description: Serious adverse events (SAEs) defined as untoward medical occurrence that at any dose: results in death, is life-threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires in subject hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event (defined as a medical event(s) that may not be immediately life-threatening or result in death or hospitalization but, may jeopardize the subject or may require intervention to prevent one of the other serious outcomes listed in the definition above.)
Time Frame: 4 months
Population: All subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab Treatment + Radiation Therapy
Number analyzed (Participants) | 22
Participants | 9

2. Secondary Outcome: Response Rate
Description: Compare tumor response rate and duration of response at unirradiated sites in patients with Stage IV melanoma with historical controls.
  Response assessed per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by physical measurement; magnetic resonance imaging (MRI); computed tomography (CT), positron emission tomography (PET)-CT; and/or X-rays:
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
Time Frame: 2 to 4 weeks after last ipilimumab dose then every 3 months +/- 2 weeks until progression of disease
Population: All subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab Treatment + Radiation Therapy
Number analyzed (Participants) | 22
Participants | 11

3. Secondary Outcome: Overall Survival
Description: Median time to overall survival was calculated using the Kaplan-Meier algorithm.
Time Frame: 2 to 4 weeks after last ipilimumab dose then every 3 months +/- 2 weeks until progression of disease
Population: All subjects
Measure: Median (Full Range); unit: weeks
Arm/Group | Ipilimumab Treatment + Radiation Therapy
Number analyzed (Participants) | 22
weeks | 107 [7 to 214]

4. Secondary Outcome: Duration of Complete Response
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.
Time Frame: 2 to 4 weeks after last ipilimumab dose then every 3 months +/- 2 weeks until progression of disease
Population: all subjects
Measure: Median (Full Range); unit: weeks
Arm/Group | Ipilimumab Treatment + Radiation Therapy
Number analyzed (Participants) | 3
weeks | 112 [60 to 139]

5. Secondary Outcome: Duration of Partial Response.
Description: Length of time between first dose of ipilimumab and a partial response according to RECIST v1.1 (see above) and immune response criteria
Time Frame: 2 to 4 weeks after last ipilimumab and then every 3 months until disease progression.
Population: all patients that did not have SAEs during treatment and did not have complete response.
Measure: Median (Full Range); unit: weeks
Arm/Group | Ipilimumab Treatment + Radiation Therapy
Number analyzed (Participants) | 3
weeks | 40 [29 to 53]

6. Secondary Outcome: Stable Disease
Description: Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements
Time Frame: 2 to 4 weeks after last ipilimumab and then every 3 months until disease progression.
Population: All patients who did not have SAEs during treatment and did not reach complete response or partial response.
Measure: Median (Full Range); unit: weeks
Arm/Group | Ipilimumab Treatment + Radiation Therapy
Number analyzed (Participants) | 5
weeks | 39 [26 to 76]

7. Secondary Outcome: Median Time to Complete Response or Partial Response
Description: Time from the first dose of ipilimumab to the first tumor measurement showing either a complete or partial response to therapy.
Time Frame: 2 to 4 weeks after last ipilimumab and then every 3 months until disease progression.
Population: All patients who had either a complete response or partial response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ipilimumab Treatment + Radiation Therapy
Number analyzed (Participants) | 6
weeks | 19 [12 to 52]

8. Secondary Outcome: Progression-free Survival (PFS)
Description: Median time to progression-free survival (PFS) was calculated using the Kaplan-Meier algorithm
Time Frame: 2 to 4 weeks after last ipilimumab and then every 3 months until disease progression.
Population: All subject who did not have SAEs during treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ipilimumab Treatment + Radiation Therapy
Number analyzed (Participants) | 20
weeks | 26 [9 to 50]

ADVERSE EVENTS:
Time Frame: Collected form first dose of study drug until the end of active follow up.
Arm/Group | Ipilimumab Treatment + Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 13/22
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab Treatment + Radiation Therapy (N=22)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Hemorrhage, CNS (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (5)
Anemia (Blood and lymphatic system disorders) | 1 (1)
dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Enteritis (Gastrointestinal disorders) | 1 (1)
INFECTION-Other: Sepsis (Infections and infestations) | 1 (1)
INFECTION-Systemic Inflammatory Response Syndrome (SIRS) (Infections and infestations) | 1 (1)
Melena (Gastrointestinal disorders) | 1 (1)
new brain lesion (Nervous system disorders) | 1 (1)
PAIN-GASTROINTESTINAL-Abdomen NOS (Gastrointestinal disorders) | 4 (6)
Vomitting (Gastrointestinal disorders) | 4 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab Treatment + Radiation Therapy (N=22)
Diarrhea (Gastrointestinal disorders) | 14 (20)
Fatigue (General disorders) | 15 (16)
Nausea (Gastrointestinal disorders) | 12 (17)
Rash: Erythema (Skin and subcutaneous tissue disorders) | 10 (13)
Vomiting (Gastrointestinal disorders) | 9 (13)

LIMITATIONS AND CAVEATS:
This study was intended to be exploratory and had a limited sample size. Our results are based on a small sample size and further research should be done to really draw firm conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes